CLINICAL TRIAL: NCT04574206
Title: Developing and Evaluating a Parent-child Intervention for Intellectually Able Children With Autism Spectrum Disorders: A Feasibility Study
Brief Title: Testing a Novel Parenting Intervention for Children With Autism
Acronym: PAREint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GRY190053860
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomised pilot study to compare a caregiver-delivered elaborative reminiscence intervention against a control intervention for children with autism spectrum disorder, aged 7-11 years. Randomisation will occur at the participant level and participants will be allocated to the trial arms using a 1:1 ratio.
Who Masked: Participant
Masking Description: The study will be single-blinded at the participant level, however if further funding is obtained then the study will be double-blinded to include blinding at the researcher level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elaborative Reminiscence (ER) (Experimental): ER is a communication strategy used between a caregiver and child to support children's cognitive and emotional development. ER involves a caregiver and child jointly reminiscing about a past event that they personally experienced, to co-create a coherent narrative that describes the event from both their perspectives. ER consists of two crucial elements, the use of elaborative language (e.g. open ended questions, contributing new information to the conversation) and specific talk focused on recollections of the past as opposed to observations of the present.
  Interventions: Behavioral: Elaborative Reminiscence (ER)
- Present Tense Talk (PTT) (Sham Comparator): PTT is an active control intervention, designed to ensure that caregivers/ guardians in this group spend a similar amount of time engaging in conversation with their children but do not use elaborative reminiscing language. The focus will be on describing activities as they are happening in real time; PTT caregivers will be asked to avoid reference future or past events .
  Interventions: Behavioral: Present Tense Talk (PTT)

INTERVENTIONS:
Behavioral: Elaborative Reminiscence (ER) — Parents will be trained to use elaborative communication techniques in conversations with their child.
  Arms: Elaborative Reminiscence (ER)
Behavioral: Present Tense Talk (PTT) — Parents will be trained to engage their children in conversations, describing activities as they are actually happening.
  Arms: Present Tense Talk (PTT)

SUMMARY:
This study will investigate the acceptability and preliminary effectiveness of training parents to use a structured communication intervention that is aimed towards helping children with autism spectrum disorder (ASD).

This intervention has demonstrated benefits for non-autistic children in known areas of difficulty found with autistic individuals. There are currently few evidence-based interventions for school-aged children with ASD who have no other language or intellectual disabilities and are educated in mainstream schools. We will evaluate the benefits of training parents to use a freely available communication technique designed to tackle underlying psychological processes crucial to later development.

DETAILED DESCRIPTION:
Over recent years a growing body of research has reported significant, beneficial effects of using an "elaborative reminiscence" (ER) intervention on a range of typically-developing child outcomes including memory language skills, emotional understanding and understanding of mind. A recently published 9- year follow-up study further indicates that these benefits are longstanding. This has prompted speculation that ER could be a beneficial intervention for children with neurodevelopmental disorders who have known difficulties in these areas. To date, no studies have assessed the benefits of using ER as an intervention for ASD.

This study aims to evaluate the feasibility, acceptability and preliminary effectiveness of training parents to use ER as an intervention for high-functioning children with ASD. This study will use a two-arm, parallel-group, randomised controlled design to compare a parent-delivered ER intervention against a control intervention (present tense talk).

Fifty parent-child dyads (comprising children with ASD and IQ >70) will be recruited from mainstream schools, specialist unit/ schools, or relevant organisations (25 dyads per trial arm). Primary outcomes will be NIHR-recognised quantitative indicators of feasibility and acceptability for the ER condition.This will include (yet is not limited to) exploring the feasibility of methods of recruiting participants, feasibility of administering outcome assessments at baseline and follow-up, feasibility of delivering the training for ER and PTT remotely (i.e. through video conferencing), the feasibility of parents delivering ER or PTT in their home setting, and the acceptability of ER to parents. Parent acceptability of ER will be assessed using a daily logbook questionnaire and post-trial interviews, based on the Theoretical Framework of Acceptability.

Secondary outcomes will be measures of clinical and functional outcomes for both experimental conditions. Descriptive measures of general intelligence, vocabulary and developmental level will be administered at baseline for both experimental conditions (ER and PTT) and used to describe the participant sample. Outcome measures for child memory, mental state understanding, and self-concept will be administered at baseline and again after 20 weeks to assess change or response to the interventions. Differences in parent reminiscing style from baseline to post-trial will be assessed for all participants to assess the success of intervention training.

On completion of follow-up outcome assessments, parents in the ER condition will be invited to participate in a single qualitative interview to evaluate the acceptability of the ER intervention and study procedures. Interviews will be based on the Theoretical Framework of Acceptability and the Necessity-Concerns Framework.

Descriptive statistics will be taken for indicators of intervention feasibility and acceptability.Comparisons between the two trial arms will be made using inferential statistical analysis for multiple outcomes, whilst adjusting for covariates.

In response to the present Covid-19 situation, this study will take place remotely. All interaction with participants (recruitment and data collection and participant testing) will use video software (e.g. Zoom, AdobeConnect, MS Teams), or online surveys (e.g. Qualtrics). Data analysis will either take place in the Autism Research Unit laboratory, located at City University of London, or remotely via a secure network.

ELIGIBILITY:
Inclusion Criteria:

Caregivers and children:

1. Must have access to a digital device capable of receiving video calls (e.g. smartphone, tablet or computer) and internet
2. Must primarily speak in English, as assessed with a pre-screening survey question.

Children only:

1. Aged 7-11 years
2. Diagnostic status i) Documented clinical diagnosis of ASD provided by caregivers or schools (e.g. a diagnostic report), OR ii) Meeting cut off for autism on the Social Communication Questionnaire (i.e. Score above or equal to 15 on SCQ)
3. Intelligence within the average range or above as measured by the Raven's Coloured Progressive Matrices (ie minimum IQ within 2 SD below the mean).
4. Developmental and linguistic levels within the average range as measured by the Vineland Adaptive Behaviour Scales (VABS-3) and the British Picture Vocabulary Scale (BPVS).

Exclusion Criteria:

Caregivers and children:

3) Must not currently be receiving care or treatment for a mental or psychiatric condition 4) Must not be currently taking part in another research study

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Trial recruitment feasibility | 20 weeks post-trial
  The number of participants who dropped out of the trial as a percentage of the total number recruited.
Feasibility of training procedures | Baseline
  Percentage of participants who demonstrate 70% or more of intervention behaviours during the training roleplay assessment.
Training enactment | Change from baseline to 20 weeks post-trial
  Change to caregiver reminiscing style ratio following training
Implementation fidelity (actual dosage) | 20 weeks post-trial
  The actual number of intervention behaviours caregivers demonstrate during conversations at post-trial.
Implementation fidelity (frequency of intervention delivery) | 20 weeks post-trial
  The mean number of intervention minutes delivered by caregivers
Intervention acceptability | 20 weeks post-trial
  A qualitative analysis (guided by the Theoretical Framework of Acceptability) of post-trial caregiver interviews to determine caregiver acceptability of the ER intervention.

SECONDARY OUTCOMES:
Memory test | Change from baseline to 20 weeks post-trial
  Change to child scores on the California Verbal Learning Test for Children (CVLT-C)
Memory elaborations | Change from baseline to 20 weeks post-trial
  Number of child memory elaborations during parent-child conversations
Mental state understanding | Change from baseline to 20 weeks post-trial
  Change to child scores on the Theory of Mind Battery
Self-concept | Change from baseline to 20 weeks post-trial
  Change to child scores on the Self-Description Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ramberg, Study Director — City, University of London
Locations (1):
- City University of London, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As this is a PhD research study, no plan nor ethical approval has yet been obtained to make IPD available to other researchers.